CLINICAL TRIAL: NCT05331534
Title: Evaluation of the Effectiveness of Eye-tracking Assisted Attentional Bias Reduction Therapy on Reducing Symptoms of Post-traumatic Stress Disorder
Brief Title: Effect of Attentional Therapy on Post-traumatic Stress Disorder
Acronym: BATRAUMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021_0860; 2022-A00224-39 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-03-21; First posted 2022-04-15 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Post-traumatic stress disorder; Attentional bias; Eye tracking; Attention Control Training
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with a PTSD receiving ACTo and prolonged exposure therapy. (Experimental)
  Interventions: Behavioral: Eye-tracking assisted attention control training (ACTo)
- patients with PTSD receiving ACT and prolonged exposure therapy. (Sham Comparator)
  Interventions: Behavioral: Attention control training (ACT)

INTERVENTIONS:
Behavioral: Eye-tracking assisted attention control training (ACTo) — ACT is made of 8 sessions of a Dot-Probe Task (DPT). The DPT is a computerized task in which two visual stimuli (one emotional stimulus and one neutral stimulus) are displayed simultaneously on the left and right side of the screen. AB towards or away from emotional stimuli is respectively inferred by faster or slower responses to detect a probe replacing an emotional stimulus than a probe replacing a neutral stimulus. In the ACT therapy, the probe replaces the negative and neutral stimuli with equal frequency.
  ACTo will combine ACT with eye tracking methodology, allowing to directly record eye movements of the participants during the task. At each trial, images will be displayed for 2s and the negative image will be replaced by the neutral image (and vice versa) if the patient continues to explore the negative image beyond the first fixation, in order to block any additional attentional engagement.
  Arms: patients with a PTSD receiving ACTo and prolonged exposure therapy.
Behavioral: Attention control training (ACT) — Patients will benefit from the ACT as described above; at each trial, images will remain on screen for 2s.
  Arms: patients with PTSD receiving ACT and prolonged exposure therapy.

SUMMARY:
Post-traumatic stress disorder (PTSD) is associated with an attentional bias towards negative stimuli, which is supposed to contribute to the development and the maintenance of the disorder. We recently showed using eye-tracking evidenced two types of AB towards negative stimuli: a "physiological AB" found both in healthy and individual with PTSD, characterized by a stronger initial attentional engagement towards negative stimuli compared to neutral stimuli, as revealed by longer first fixation duration dwell time on negative pictures than on neutral pictures; a "pathological bias" observed only in individuals with PTSD and characterized by an heightened sustained attention towards negative stimuli once detected, which further increases with prolonged exposure. The present study aimed at assessing the effectiveness of an eye-tracking assisted attentional bias reduction therapy, targeting specifically the pathological bias on the reduction of PTSD symptoms

ELIGIBILITY:
Inclusion Criteria:

* Understanding and able to express themselves in French
* Giving informed consent, by dating and signing the study participation form
* Having health insurance coverage
* Normal or corrected to normal vision and hearing
* DSM-5 PTSD criteria, assessed using the CAPS and PCL-5

Exclusion Criteria:

* Minors or adults under guardianship, under judicial protection, persons deprived of liberty
* Pregnant or breastfeeding women
* Refusal to participate after being clearly and fairly informed about the study
* Sensory, visual or auditory incapacity to participate in the study
* Personal history of neurological disorder or current neurological disorder
* Use of drugs other than tobacco and alcohol
* Alcohol use on the day of experimentation
* Personal history of psychiatric disorders or current psychiatric disorders other than anxiety, depressive, or trauma and stress disorders assessed at clinical interview and with MINI
* Personal history of multiple trauma in childhood
* Psychotropic medication treatment not stabilized over the past 4 weeks
* MOCA < 26
* Contraindication to prolonged exposure therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2028-02-02 (Estimated); Study Completion 2029-02-02 (Estimated)

PRIMARY OUTCOMES:
PTSD symptomatology assessed using the Clinician-Administered PTSD Scale (CAPS) score. | Before and after ACTo or ACT treatment: at day 1 and 1 month after inclusion
  The CAPS-5 is a 30-item structured interview corresponding to the DSM-5 diagnosis for PTSD. The CAPS-5 combines information about frequency and intensity of an item into a single severity rating (range 0-4). CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms. Similarly, CAPS-5 symptom cluster severity scores are calculated by summing the individual item severity scores for symptoms corresponding to a given DSM-5 cluster. Higher scores thus correspond to higher severity of PTSD symptoms.

SECONDARY OUTCOMES:
AB will be assessed in both groups by measuring the total fixation time on negative versus neutral images in a dot-probe task with eye tracking | Before and after ACTo or ACT treatment: at day 1 and 1 month after inclusion
Calculation of correlation coefficients between pre- and post-treatment differences in AB and PTSD | Before and after ACTo or ACT treatment: at day 1 and 1 month after inclusion
  AB will be measured by total fixation time on negative versus neutral images in a dot-probe task with eye tracking; and psychotraumatic symptomatology will be measured by the Clinician-Administered PTSD Scale (CAPS).
The number of sessions of prolonged exposure therapy required to achieve a score below the clinical cut-off at the PTSD Checklist for DSM-5 (PCL5) (<33/80) | Before each prolonged exposure therapy session: 1 month after inclusion, during 3 months on average
  The PTSD Checklist for DSM-5 (PCL5) is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items. Higher scores indicate more symptoms of PTSD. A score above 32 suggests a probable PTSD.
Follow-up on psychotraumatic symptomatology will be assessed using the Clinician-Administered PTSD Scale (CAPS) score | One month after prolonged exposure therapy treatment, up to 6 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Vaiva, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Fontan 2, Lille, France

IPD SHARING:
Plan to Share IPD: No